CLINICAL TRIAL: NCT05132452
Title: The Test of Mastication and Swallowing Solids and the Timed Water Swallow Test: Reliability, Associations, Age and Gender Effects, and Normative Data
Brief Title: The Test of Mastication and Swallowing Solids and the Timed Water Swallow Test
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Oshrat Sella, Principal Investigator, University of Haifa
Other Study IDs: 1012
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Healthy Aging; Gender; Swallowing Disorder
MeSH Terms: conditions — Coitus; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- adults living in the community: Healthy community dwelling participants, aged 20 year old and above, without dysphagia.
  Interventions: Diagnostic Test: The Test of Mastication and Swallowing Solids (TOMASS) and the Timed Water Swallow Test (TWST)

INTERVENTIONS:
Diagnostic Test: The Test of Mastication and Swallowing Solids (TOMASS) and the Timed Water Swallow Test (TWST) — Participants swallowed one cracker for the TOMASS. They swallowed 150 mL of water for the TWST.

SUMMARY:
This study aimed to gather more information regarding two clinically relevant tests: The Test of Mastication and Swallowing Solids (TOMASS) and the Timed Water Swallow Test (TWST). Both tests can be used clinically as part of swallowing disorders evaluation.

The aims of the study were to assess the reliability of the two tests, to document the effects of age and gender on the outcome measures of the TOMASS and TWST and to explore the relationship between participants' function in the two tests. To do that, 298 healthy participants were included. All of them did not have dysphagia. Most of them were elderly.

DETAILED DESCRIPTION:
Background: Quantitative measures of swallowing function can increase accuracy, reliability, and improve clinical decision making. The Test of Mastication and Swallowing Solids (TOMASS) and the Timed Water Swallow Test (TWST) are functional tests of swallowing that provide quantitative results.

Objectives: To explore the relationship between TOMASS and TWST; evaluate test-retest and interrater reliability; explore age and gender effects; and to gather normative data.

Methods: Healthy community dwelling participants (n = 298, ≥20 years old) were recruited. Of those, 126 were included in the reliability study. Participants completed the TWST and TOMASS.

ELIGIBILITY:
Inclusion Criteria:

* all participants were eligible to participate if they were over 20 years of age, with no known medical history of dysphagia, had an SDQ score of less than 11, indicating no suspicion for dysphagia, were able to give a written informed consent, and could follow simple verbal instructions. In addition, all participants indicated that they do not avoid eating crackers due to swallowing disorders or allergies.

Exclusion Criteria:

* SDQ over 11 or medically reported dysphagia not eating crackers due to swallowing difficulty allergy to gluten

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects living in the community
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
duration | one-off assessment
  length of time required to complete the task
swallows | one-off assessment
  number of swallows required to complete the task
bites | one-off assessment
  number of bites required to eat the cracker
masticatory cycles | one-off assessment
  number of masticatory cycles required to eat the cracker
volume | one-off assessment
  the amount of water swallowed

CONTACTS AND LOCATIONS:
Overall Officials: oshrat sella, PhD, Principal Investigator — University of Haifa

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Sarve AR, Krishnamurthy R, Balasubramanium RK. The timed water test of swallowing: Reliability, validity, and normative data from Indian population. Int J Health Sci (Qassim). 2021 Mar-Apr;15(2):14-20. PMID 33708040
- [Result] Athukorala RP, Jones RD, Sella O, Huckabee ML. Skill training for swallowing rehabilitation in patients with Parkinson's disease. Arch Phys Med Rehabil. 2014 Jul;95(7):1374-82. doi: 10.1016/j.apmr.2014.03.001. Epub 2014 May 9. PMID 24816250
- [Result] Huckabee ML, McIntosh T, Fuller L, Curry M, Thomas P, Walshe M, McCague E, Battel I, Nogueira D, Frank U, van den Engel-Hoek L, Sella-Weiss O. The Test of Masticating and Swallowing Solids (TOMASS): reliability, validity and international normative data. Int J Lang Commun Disord. 2018 Jan;53(1):144-156. doi: 10.1111/1460-6984.12332. Epub 2017 Jul 5. PMID 28677236
- [Result] Krishnamurthy R, Kothari S, Balasubramanium RK, Huckabee ML. The Test of Masticating and Swallowing Solids (TOMASS): Normative data for the adult Indian population. Data Brief. 2021 Mar 18;35:106958. doi: 10.1016/j.dib.2021.106958. eCollection 2021 Apr. PMID 33850987
- [Result] Hughes TA, Wiles CM. Clinical measurement of swallowing in health and in neurogenic dysphagia. QJM. 1996 Feb;89(2):109-16. doi: 10.1093/qjmed/89.2.109. PMID 8729551